CLINICAL TRIAL: NCT04632069
Title: N-acetylcysteine Plus Transcutaneous Vagus Nerve Stimulation in Infants of Diabetic Mothers Who Fail Oral Feeding
Brief Title: NAC +taVNS in IDM Who Are Poor Oral Feeders
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Dorothea D. Jenkins, Professor of Pediatrics, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103800; P20GM109040 (NIH)
Record Dates: First submitted 2020-11-12; First posted 2020-11-17 (Actual); Results first posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Infant of Diabetic Mother; Oxidative Stress; Vagus Nerve Stimulation; Feeding Disorders
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Acetylcysteine; Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: We will obtain parental consent, and then administer NAC 100mg/kg loading dose, followed by 75mg/kg q 6h via nasogastric tube, started 4 days prior to taVNS-paired feeding and continued for a total of 14 days. We will perform pharmacokinetics of oral NAC, and MRIs prior to, after 3-4 days of NAC, and after taVNS treatment period.
Masking Description: Co-investigator analyzing MRI data will be blinded to timing of MRI scan and dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- NAC + taVNS (Experimental): NAC will be given via nasogastric tube (n,g.) 100mg/kg loading dose, then 75mg/kg/dose n.g. q 6h, administered 1h before a feed, for a total of 14 days. taVNS will be administered to left ear during active sucking with 2 daily feedings starting after 4 days of NAC, continuing for 10 days.
  Interventions: Combination Product: N acetyl cysteine + vagus nerve stimulation

INTERVENTIONS:
Combination Product: N acetyl cysteine + vagus nerve stimulation — NAC x 14 days, taVNS x 10 days
  Other Names: NAC, Acetadote, taVNS

SUMMARY:
Infants of diabetic mothers who are failing to learn oral feeding by term age equivalence have greater CNS oxidative stress, which interact to predict poor neuroplasticity response to transcutaneous vagus nerve stimulation paired with oral feeding. We propose treating the oxidative stress in IDM infants prior to initiating taVNS, with an FDA-approved antioxidant (N-acetylcysteine, NAC) to improve CNS oxidative stress, which in turn regulates expression of many genes including BDNF, that may enhance motor learning.

DETAILED DESCRIPTION:
Our group has recently conducted a first-in-infants pilot trial of pairing transcutaneous auricular vagus nerve stimulation (taVNS) with feeding to assist learning oromotor skills. We are enrolling preterm and HIE infants who are failing to learn oral feeds and clinically determined to need a G-tube. In preliminary data, taVNS paired with one or two daily feedings for 2 weeks resulted in 50% of infants attaining full feeds and avoiding G-tube.

A notable number of non-responders were infants of diabetic mothers (IDM) exposed to poor glucose control during pregnancy, all of whom required a G-tube. Uncontrolled maternal hyperglycemia is associated with increased systemic and neuro-inflammation, CNS oxidative stress, DNA damage, and worse neonatal outcomes compared to infants of euglycemic mothers. In neonatal animal models, hyperglycemia has been shown to decrease BDNF, alter long-term synaptogenesis and hippocampal neurochemistry, with ongoing CNS oxidative stress and inhibition of the cortical neuronal plasticity required for learning. In our pilot trial of taVNS-paired feeding, CNS glutathione concentrations (GSH), a MR spectroscopy (MRS) marker of oxidative stress, had significant interaction with IDM in predicting outcome, strongly suggesting that ongoing CNS oxidative stress contributes to neuropathology in IDMs failing oral feeding.

NAC is an FDA-approved antioxidant that is safe and crosses the blood brain barrier, increasing CNS GSH. NAC reduces CNS oxidative stress, enhances learning and provides a neuroprotective effect after brain injury in our and others neonatal HI and neuroinflammatory animal models. Both GSH and BDNF enhance neuroplasticity. Therefore, we hypothesize that pre-treatment with NAC in IDMs who are failing oral feeding, followed by taVNS-paired feeding, will decrease oxidative stress induced by maternal hyperglycemia and IDM-associated brain injury, and increase response to taVNS-paired feeding rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Infants of diabetic mothers who are failing oral feeding, >39weeks gestation at enrollment, who are clinically stable, on minimal respiratory support (nasal cannula or room air), and clinical team has determined are G-tube candidates

Exclusion Criteria:

* Unstable infants or those requiring positive pressure respiratory support
* Infants <39 weeks gestation at enrollment
* Major unrepaired congenital anomalies or anomalies that limit feeding volumes
* Infants with cardiomyopathy
* Repeated episodes of autonomic instability (apnea/ bradycardia) not self resolving

Ages: 3 Weeks to 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothea Jenkins, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
will share de-identified data after publication of results
Supporting Information: Study Protocol
Time Frame: after publication of results
Access Criteria: written request of PI

REFERENCES:
- [Background] Badran BW, Jenkins DD, Cook D, Thompson S, Dancy M, DeVries WH, Mappin G, Summers P, Bikson M, George MS. Transcutaneous Auricular Vagus Nerve Stimulation-Paired Rehabilitation for Oromotor Feeding Problems in Newborns: An Open-Label Pilot Study. Front Hum Neurosci. 2020 Mar 18;14:77. doi: 10.3389/fnhum.2020.00077. eCollection 2020. PMID 32256328
- [Background] Badran BW, Jenkins DD, DeVries WH, Dancy M, Summers PM, Mappin GM, Bernstein H, Bikson M, Coker-Bolt P, George MS. Transcutaneous auricular vagus nerve stimulation (taVNS) for improving oromotor function in newborns. Brain Stimul. 2018 Sep-Oct;11(5):1198-1200. doi: 10.1016/j.brs.2018.06.009. Epub 2018 Jun 30. No abstract available. PMID 30146041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from 8.12.21 to 3.1.23 in the Neonatal intensive care unit of the Medical University of South Carolina
Groups:
- NAC + taVNS: NAC will be given via nasogastric tube (n.g.) 75mg/kg/dose or 100mg/kg/dose n.g. q 6h, administered 1h before a feed, for a total of 14 days. taVNS will be administered to left ear during active sucking with 2 daily feedings starting after 4 days of NAC, continuing for 10 days.
  N acetyl cysteine + vagus nerve stimulation: NAC x 14 days, taVNS x 10 days
Period: Overall Study
Arm/Group | NAC + taVNS
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- NAC + taVNS: NAC will be given via nasogastric tube (n,g.) 75mg/kg/dose or 100mg/kg n.g. q 6h, administered 1h before a feed, for a total of 14 days. taVNS will be administered to left ear during active sucking with 2 daily feedings starting after 4 days of NAC, continuing for 14 days.
  N acetyl cysteine + vagus nerve stimulation: NAC x 14 days, taVNS x 14days
Arm/Group | NAC + taVNS
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: weeks post menstrual age] — age an enrollment
  weeks post menstrual age | 41.1 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants] — male/female
  Participants
    Female | 4
    Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — hispanic or nonhispanic
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 9
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — USA, Charleston, SC
  participants
    United States | 10
mean daily oral feeding volume of formula or breast milk [Mean (Standard Deviation); unit: ml/kg/day] — mean daily oral feeding volume averaged over 14 days
  ml/kg/day | 47 (29)

OUTCOME MEASURES:

1. Primary Outcome: Daily Oral Feeding Volumes : Difference in Mean Increase
Description: Difference in the Mean daily change in oral feeding volume(reported in in ml/kg/d) from Day 1-18 days of NAC+taVNS treatment minus Days -14 to 0 (baseline)
Time Frame: Day -14 to 0, Day 1 to 18
Population: infants of diabetic mothers failing oral feeds in G-tube discussions
Measure: Mean (Standard Deviation); unit: ml/kg/day po daily change
Groups:
- NAC + taVNS: NAC will be given via nasogastric tube (n,g.) 75 or 100mg/kg n.g. q 6h, administered 1h before a feed, for a total of 14 days. taVNS will be administered to left ear during active sucking with 2 daily feedings starting after 4 days of NAC, continuing for 14 days.
  N acetyl cysteine + vagus nerve stimulation: NAC x 14 days, taVNS x 14 days
Arm/Group | NAC + taVNS
Number analyzed (Participants) | 10
ml/kg/day po daily change | 2.1 (0.4)
Statistical Analysis 1: Comparison: NAC + taVNS; Daily change in po feeding volumes expressed as po ml/kg/d [reported as the mean daily change from Day 1 to 18 during NAC/NAC+taVNS minus baseline mean daily change Day -14 to day 0 (before treatment)] Null hypothesis: there will be no significant difference in daily change in po feeding volume (ml/kg/d) from baseline to during treatment Power analysis: Estimated +0.2 ml/kg/d before taVNS, and +3ml/kg/d during the 18days of NAC+taVNS treatment, requiring 10 infants with power of 80%, a=0.05; Test type: Superiority; p = 0.009, Regression, Linear; repeated measures linear regression: time periods: -14 to Day 0, Day 1-18(independent variable); daily po volumes (Dependent Variable); Mean Difference (Final Values) = 2.1, Standard Deviation 0.4

2. Secondary Outcome: Metabolite Concentrations in Basal Ganglia
Description: Change in [GSH] by MRS from baseline to day 4 of NAC
Time Frame: baseline to 4 days
Population: participants with adequate MRS spectra for analysis
Measure: Mean (Standard Deviation); unit: mM
Groups:
- NAC + taVNS: NAC will be given via nasogastric tube (n,g.) 75 or 100mg/kg n.g. q 6h, administered 1h before a feed, for a total of 14 days. taVNS will be administered to left ear during active sucking with 2 daily feedings starting after 4 days of NAC, continuing for 14days.
  N acetyl cysteine + vagus nerve stimulation: NAC x 14 days, taVNS x 14 days
Arm/Group | NAC + taVNS
Number analyzed (Participants) | 8
mM | 0.13 (.08)
Statistical Analysis 1: Comparison: NAC + taVNS; [GSH] at baseline compared with [GSH] at day 4 of NAC- by paired t-test in which each participant's [GSH] is compared at 2 time points Null hypothesis: the [GSH] in the basal ganglia will be no different after Day 4 of NAC than [GSH] at baseline Power calculation:With 80% power, alpha of 0.05, we would need 7 patients to show a significant change in basal ganglia [GSH] of 0.14 +/- 0.13mM from baseline to Day 4 of NAC (paired t-test); Test type: Superiority; p = 0.01, t-test, 2 sided; paired t-test; Mean Difference (Final Values) = 0.13, Standard Deviation .08 — mean difference between [GSH] Day 4 of NAC and [GSH] at baseline

ADVERSE EVENTS:
Time Frame: 36 days
Description: bradycardia defined as heart rate <80beats per minute for > 5 seconds; emesis
Arm/Group | NAC + taVNS
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAC + taVNS (N=10)
bradycardia (Cardiac disorders) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NAC + taVNS (N=10)
emesis per day (Gastrointestinal disorders) | 2 (2) — emesis after NAC administration with dilution 1:2 with sterile water. no further emesis with dilution 1:3

LIMITATIONS AND CAVEATS:
small numbers in phase I trial; non concurrent control group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT04632069/Prot_SAP_001.pdf
  • Informed Consent Form (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/69/NCT04632069/ICF_000.pdf